CLINICAL TRIAL: NCT00877396
Title: Does Vaccinating Health Hutterite Children Against Influenza Prevent Influenza in Other Hutterite Colony Members: A Randomized Cluster Trial
Brief Title: Hutterite Influenza Prevention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mark Loeb, Study Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCT 88113
Record Dates: First submitted 2009-01-22; First posted 2009-04-07 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza (Experimental): Inactivated Influenza vaccination
  Interventions: Biological: Influenza vaccination
- Control (Placebo Comparator): Hepatitis A vaccine
  Interventions: Biological: Hepatitis A Vaccine

INTERVENTIONS:
Biological: Influenza vaccination — Influenza vaccination- 0.5 mL. Children under 9 who have never received a influenza vaccine will receive a 2nd dose (0.5 mL) 4 weeks later.
  Other Names: Vaxigrip by Sanofi Pasteur
  Arms: Influenza
Biological: Hepatitis A Vaccine — Hepatitis vaccination- 0.5 mL. Children under 9 who have never received a influenza vaccine will receive a 2nd dose ( saline- 0.5 mL) 4 weeks later.
  Other Names: Avaxim Pediatric by Sanofi Pasteur
  Arms: Control

SUMMARY:
The goal of this randomized clinical trial is to determine whether immunizing children in Hutterite colonies with inactivated influenza vaccine can prevent influenza and its complications in other colony members. Furthermore, the study will assess the indirect benefit to Hutterites at high risk of complications. The study is a blinded, cluster randomized controlled trial among Hutterite colonies to test the hypothesis that high immunization rates (>70%) of healthy children with inactivated influenza vaccine reduces transmission of influenza to other colony members. Randomization of these homogeneous, moderately sized colonies where there is regular spread facilitated by a communal lifestyle, but limited re-introduction because of relative isolation from outside community, represents a unique opportunity to test the hypothesis of indirect benefit under close to ideal conditions. The primary outcome will be laboratory-confirmed influenza. Secondary outcomes include influenza-like illness, otitis media, physician visits, antimicrobial prescriptions, absenteeism, lower respiratory tract infection, hospitalizations, and death.

DETAILED DESCRIPTION:
Colonies will be enrolled in September 2008.

Healthy Hutterite Children will be vaccinated in October, in each year of the study (2008, 2009, & 2010)

Influenza Surveillance phase will begin around December-January of each year.

* All study outcomes will be collected during the Surveillance phase of the study from Dec to June for 3 years.
* Outcomes will be collected when research nurses visit the colonies. A research nurse will visit enrolled colonies twice a week during the surveillance phase and review study diaries and obtain swabs from participants with symptoms of influenza.

ELIGIBILITY:
Group A:

Inclusion Criteria:

* Hutterites other than the healthy children who will be immunized. Although this category as a whole will be used to assess indirect benefit of the vaccine in the main analysis, Hutterites at high risk for influenza complications within this category will be assessed in a separate analysis. These are defined as anyone in one or more of the following groups:
* individuals aged ≥ 65 years
* children 23 months of age or less
* anyone with ≥ 1 of the following conditions severe enough to require regular medical follow-up or hospital care:

  * chronic cardiac or pulmonary disorders (including bronchopulmonary dysplasia, cystic fibrosis, and asthma)
  * diabetes mellitus and other metabolic diseases
  * cancer
  * immunodeficiency
  * immunosuppression (due to underlying disease and/or therapy)
  * renal disease
  * anemia
  * hemoglobinopathy
  * any condition that can compromise respiratory function or the handling of respiratory secretions or that can increase the risk of aspiration.

Exclusion Criteria:

* There are no exclusion criteria for this category of participants.

Group B:

Inclusion Criteria:

* Healthy children aged 36 months to 15 years who will be immunized as part of the intervention.

Exclusion Criteria:

* Anaphylactic reaction to a previous dose of influenza vaccine
* Anaphylactic reaction to hepatitis A vaccine
* Anaphylactic reaction to neomycin
* Known IgE-mediated hypersensitivity to eggs manifested as hives
* Swelling of the mouth and throat, difficulty in breathing, hypotension, or shock
* Guillain-Barré syndrome within eight weeks of a previous influenza vaccine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4771 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
laboratory-confirmed influenza infection | Dec to June each year for 3 years

SECONDARY OUTCOMES:
Influenza like illness | Dec to June each year for 3 years
Physician diagnosed otitis media | Dec to June each year for 3 years
School or work related absenteeism | Dec to June each year for 3 years
Physician visits for respiratory illness | Dec to June each year for 3 years
Lower respiratory infection or pneumonia | Dec to June each year for 3 years
Hospitalizations for LRTI or pneumonia | Dec to June each year for 3 years
All cause hospitalizations | Dec to June each year for 3 years
Deaths due to LRTI or pneumonia | Dec to June each year for 3 years
All-cause deaths | Dec to June each year for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD, Principal Investigator — McMaster University

REFERENCES:
- [Derived] Wang B, Russell ML, Moss L, Fonseca K, Earn DJ, Aoki F, Horsman G, Caeseele PV, Chokani K, Vooght M, Babiuk L, Webby R, Walter SD, Loeb M. Effect of Influenza Vaccination of Children on Infection Rate in Hutterite Communities: Follow-Up Study of a Randomized Trial. PLoS One. 2016 Dec 15;11(12):e0167281. doi: 10.1371/journal.pone.0167281. eCollection 2016. PMID 27977707
- [Derived] Loeb M, Russell ML, Fonseca K, Webby R, Walter SD. Comparison of multiple estimates of efficacy for influenza vaccine. Vaccine. 2011 Dec 9;30(1):1-4. doi: 10.1016/j.vaccine.2011.10.069. Epub 2011 Nov 7. PMID 22098676
- [Derived] Loeb M, Russell ML, Moss L, Fonseca K, Fox J, Earn DJ, Aoki F, Horsman G, Van Caeseele P, Chokani K, Vooght M, Babiuk L, Webby R, Walter SD. Effect of influenza vaccination of children on infection rates in Hutterite communities: a randomized trial. JAMA. 2010 Mar 10;303(10):943-50. doi: 10.1001/jama.2010.250. PMID 20215608